CLINICAL TRIAL: NCT04358406
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Proof-Of-Concept Study To Evaluate Efficacy And Safety Of Recombinant Human Plasma Gelsolin (Rhu-pGSN) Added To Standard Of Care In Subjects With Severe Covid-19 Pneumonia
Brief Title: Rhu-pGSN for Severe Covid-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioAegis Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTI-202
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Results first posted 2023-02-09 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-09

CONDITIONS: Sars-CoV2
Keywords: COVID-19; Pneumonia; Severe; Cytokine storm
MeSH Terms: conditions — COVID-19; Pneumonia; Lymphoma, Follicular; Cytokine Release Syndrome | interventions — Gelsolin

STUDY DESIGN:
Intervention Model Description: Randomized, blinded, placebo controlled interventional
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment blinded to all but unblinded pharmacist
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Normal saline in matched volume to treatment arm. Undistinguishable in syringe.
  Interventions: Other: Placebo
- Rhu-pGSN (Active Comparator): Recombinant human plasma gelsolin reconstituted for slow bolus injection.
  Interventions: Drug: Recombinant human plasma gelsolin (Rhu-pGSN)

INTERVENTIONS:
Drug: Recombinant human plasma gelsolin (Rhu-pGSN) — Intravenous administration of rhu-pGSN at 12 mg/kg, 3 doses
  Other Names: gelsolin
  Arms: Rhu-pGSN
Other: Placebo — Normal saline in matched volume to treatment arm. Undistinguishable in syringe.
  Arms: Placebo

SUMMARY:
Study Objectives:

Primary

* To assess the efficacy (survival without organ failure on Day 14) of three doses of rhu-pGSN administered intravenously (IV) plus standard of care (SOC) to hospitalized subjects with a primary diagnosis of COVID-19 pneumonia and a severity score of 4, 5 or 6 on the World Health Organization (WHO) 9-point severity scale
* To evaluate the safety and tolerability of three IV doses of rhu-pGSN administered to hospitalized subjects with a primary diagnosis of COVID-19 pneumonia and a severity score of 4, 5, or 6 on the WHO 9-point severity scale

Secondary

* To further assess the efficacy of IV administered rhu-pGSN
* To assess changes in WHO 9-point severity score for SOC with or without rhu-pGSN
* To evaluate the effect of administered rhu-pGSN on survival rates
* To assess the relationship of pGSN levels (and other biomarkers) at baseline with clinical outcomes
* [OPTIONAL] To follow the pharmacokinetics (PK) of administered rhu-pGSN

Immunogenicity

• To investigate the development of antibodies against rhu-pGSN post-treatment

DETAILED DESCRIPTION:
Efficacy and safety of IV rhu-pGSN on top of SOC will be evaluated initially in 60 participants representative of the drug target population: high-risk subjects with acute severe pneumonia due to COVID-19. The rhu-pGSN dose will be based on actual body weight given at 12 mg/kg. Three doses will be given at 0, 12 and 24 hours intervals promptly after enrollment by IV infusion through a 0.2 µm filter. Participants will be randomized 1:1 rhu-pGSN or placebo. Interim safety analyses will be conducted after enrollment of 12, 24, 36, and 48 patients.

The primary efficacy outcome will be the proportion of patients surviving on Day 14 without mechanical ventilation, vasopressors or dialysis. Secondary efficacy outcomes will include: daily change in 9-point WHO severity score through at least Day 14; all-cause mortality at Days 28 and 90; time to death (Kaplan-Meier survival analysis); proportion of subjects alive on Days 7, 28, 60, and 90 without: ongoing use of vasopressors, ongoing intubation/mechanical ventilation, ongoing residence in an intensive care unit (ICU), new ongoing need for dialysis/renal replacement therapy; proportion of subjects discharged to home or immediate prior residence by Day 28; days on the ventilator; length of stay in hospital and in ICU and re-admission to an acute-care hospital up to Day 90. Safety of administration of rhu-pGSN at the indicated dosage will also be evaluated.

Baseline and sequential levels of pGSN and inflammatory biomarkers will be measured. On days 1, 28, and 90, immunogenicity due to the formation of anti-pGSN antibodies will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with laboratory-confirmed (RT-PCR+) or highly suspected (compatible with at least bilobar lung involvement without another plausible diagnosis) COVID-19
* Weight ≤100 kg
* Within 24 hours of reaching a WHO severity score of 4-6 either:

  * At admission
  * While already hospitalized
* Informed consent obtained from subject/next of kin/legal proxy
* Primary admitting diagnosis of pneumonia supported by a compatible clinical presentation with a documented infiltrate consistent with pneumonia on chest radiograph or CT as assessed by the admitting emergency-department (ED), clinic, or ward physician or equivalent caregiver
* Recommended (not mandatory) guidance/discretionary criteria defining patients with pneumonia satisfying all 4 categories below:

  * At least 2 symptoms: difficulty breathing, cough, production of purulent sputum, or chest pain
  * At least 2 vital sign abnormalities: fever, tachycardia, or tachypnea (thresholds -- fever: oral or core temperature >100.4 °F [38 °C]; heart rate >100 beats/min; respiratory rate >24/min)
  * At least one finding of other clinical signs and laboratory abnormalities: hypoxemia (O2 saturation <90%), clinical evidence of pulmonary consolidation, or leukocytosis or leukopenia
  * Chest imaging or CT showing new (or presumed new or worsening) pulmonary infiltrates

    * Principal investigator to note radiologic findings in the electronic case report form (eCRF)
    * Radiology report to be placed in the eCRF
    * A copy of the radiograph attached to be saved for review
* A hyperinflammatory status (defined by increased ferritin ≥500 µg/L, D-dimer ≥1000 ng/mL, or C-reactive protein (CRP) ≥75 mg/L)
* During the course of the study starting at screening and for at least 6 months after their final study treatment:

  * Female subjects of childbearing potential must agree to use 2 medically accepted birth control methods
  * Male subjects with a partner who might become pregnant must agree to use reliable forms of contraception (i.e., vasectomy, abstinence), or an acceptable method of birth control must be used by the partner
  * All subjects must agree not to donate sperm or eggs (ovocytes)

Exclusion Criteria:

* A negative RT-PCR test for COVID-19 during the evaluation of the present illness
* Extracorporeal membrane oxygenation (ECMO)
* Pregnant or lactating women
* Active underlying cancer treated with systemic chemotherapy or radiation therapy during the last 30 days
* Transplantation of hematopoietic or solid organs
* Chronic mechanical ventilation or dialysis
* Otherwise unsuitable for study participation because of chronic, severe, end-stage, and life-limiting underlying disease unrelated to COVID-19 likely to interfere with management and assessment of acute pneumonia, only comfort or limited (non-aggressive) care is to be given, or life expectancy <6 months unrelated to acute COVID infection in the opinion of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J DiNubile, MD, Study Director — BioAegis Therapeutics Inc.
Locations (3):
- Spitalul Clinic de Boli Infecţioase şi Pneumoftiziologie, Timișoara, Romania
- Spain (2):
  - Sant Joan de Reus SAM University Hospital, Reus
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Rhu-pGSN
Started (Randomized) | 33 | 31
Randomized | 33 | 31
Treated | 31 | 30
Completed | 27 | 27
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rhu-pGSN | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 78] | 64 [34 to 80] | 64 [34 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 19 | 16 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 28 | 27 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 2 | 1 | 3
  Spain | 29 | 29 | 58
World Health Organization (WHO) Severity Scale [Count of Participants; unit: Participants]
  WHO Severity 4: Oxygen by Mask or Nasal Cannula; Less severe than WHO 5. | 27 | 27 | 54
  WHO Severity 5: Noninvasive ventilation (CPAP or BiPAP) or high-flow oxygen; More severe than WHO 4 | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Proportion of Subjects Alive Not on Vasopressors, Mechanical Ventilator, or Dialysis
Description: Number and percentage of subjects alive on Day 14 without ongoing use of vasopressors, ongoing intubation/mechanical ventilation, or new/ongoing need for dialysis/RRT. Subjects who discontinued from the study early or whose survival status was inconclusive on Day 14 were considered as a failure (Not Alive).
Time Frame: Day 14
Population: Full Analysis Set: All randomized and treated with at least 1 dose of study therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
participants | 27 | 25
Statistical Analysis 1: Comparison: Placebo vs Rhu-pGSN; Test type: Superiority; p > 0.05, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Rhu-pGSN; Test type: Superiority; p > 0.1, Chi-squared

2. Primary Outcome: Safety: Number of Subjects With SAEs
Description: Number of subjects with SAEs during the study
Time Frame: Day 1 through Day 90
Population: Full Analysis Set: All randomized and treated with at least 1 dose of study therapy
Measure: Number; unit: participants
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
participants | 8 | 5

3. Secondary Outcome: Efficacy: All Cause Mortality Rate at Day 90
Description: All cause mortality rate using Kaplan-Meier survival analysis
Time Frame: Day 90
Population: Full Analysis Set: All randomized and treated with at least 1 dose of study drug
Measure: Number; unit: participants
Groups:
- Placebo: Normal saline in matched volume to treatment arm. Indistinguishable in syringe.
  Placebo: Normal saline in matched volume to treatment arm. Indistinguishable in syringe.
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
participants | 2 | 2

4. Secondary Outcome: Safety and Tolerability: Proportion of Subjects With Adverse Events (AEs)
Description: Proportion of subjects with adverse events (AEs) graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: Continuous through Day 28
Population: Full Analysis Set (all randomized and treated (At least 1 dose) subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
Participants | 16 | 16

5. Secondary Outcome: Immunogenicity: Subjects With Rhu-pGSN Antibodies
Description: Number of subjects with rhu-pGSN antibodies at Day 28
Time Frame: Day 28
Population: Full analysis set (not all tested for anti-drug antibodies at all time points on days 1, 28, and 90)
Measure: Number; unit: participants with anti-drug antibodies
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
participants with anti-drug antibodies | 7 | 7

6. Secondary Outcome: Efficacy: Alive Without Support at Day 90
Description: Number of subjects Alive without organ support at Day 90
Time Frame: Day 90
Population: Full Analysis Set: All randomized and treated with at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
participants | 28 | 25

7. Secondary Outcome: Safety and Tolerability: Proportion of Subjects With Drug-related Adverse Events (AEs)
Description: Proportion of subjects with drug-related adverse events (AEs) graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: Continuous through Day 14
Population: Full Analysis Set (all randomized and treated (At least 1 dose) subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
Participants | 0 | 1

8. Secondary Outcome: Number of Subjects Alive Without Organ Support at Day 90
Description: number of subjects alive and without organ support at the Day 90 visit
Time Frame: Through Day 90
Population: full analysis set (all treated subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Rhu-pGSN
Number analyzed (Participants) | 31 | 30
Participants | 28 | 25

ADVERSE EVENTS:
Time Frame: Entire 90 day study period
Arm/Group | Placebo | Rhu-pGSN
All-Cause Mortality (participants affected / at risk) | 2/31 | 2/30
Serious Adverse Events (participants affected / at risk) | 8/31 | 5/30
Other Adverse Events (participants affected / at risk) | 16/31 | 16/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Rhu-pGSN (N=30)
Severe acute respiratory syndrome (Infections and infestations) | 2 | 2
COVID 19 Pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
COVID 19 (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Superinfection bacterial (Infections and infestations) | 1 | 0
Acute Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diarrhoea (Eye disorders) | 0 | 1
Death (General disorders) | 0 | 1
Oxygen Saturation Decreased (Investigations) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Hemodynamic instability (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Rhu-pGSN (N=30)
SARS COV2 (Infections and infestations) | 2 | 2
COVID 19 (Infections and infestations) | 1 | 2
Transaminase Increase (Investigations) | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 3 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Hypertension (Vascular disorders) | 3 | 1
Acute Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT04358406/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT04358406/SAP_001.pdf